CLINICAL TRIAL: NCT06287723
Title: French Assessment of Minimal Residual Disease by Liquid Biopsies in Colorectal With Liver Metastasis Patients
Brief Title: French Assessment of MRD by Liquid Biopsies in Colorectal With Liver Metastasis Patients (FRENCH.MRD.CRLM)
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0297
Record Dates: First submitted 2024-02-08; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Liver Metastases; Stage IV Colorectal Cancer; Minimal Residual Disease; Liquid Biopsy; ctDNA
Keywords: Stage IV colorectal cancer; Minimal Residual Disease; Liquid biopsy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm, Residual | interventions — Blood Specimen Collection; Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA analysis NGS on tumor specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage IV colorectal liver metastasis patients: Stage IV colorectal liver metastasis patients treated with curative intent
  Interventions: Biological: Blood sample/Liquid biopsy

INTERVENTIONS:
Biological: Blood sample/Liquid biopsy — ctDNA analysis

SUMMARY:
Improving personalized cancer treatments and finding the best strategies to treat each patient relies on using new diagnostic technologies. Currently, for colorectal cancer, the methods used to decide who gets additional post-surgery treatment are suboptimal. Some patients get too much treatment, while others do not get enough.

There is a new way to explore if there is any cancer left in a patient's body using circulating tumor DNA (ctDNA) detected in blood samples. This can help decide who needs more treatment after surgery. Even though many tests have been developed, it has yet to be determined which test performs best at relevant time points.

The GUIDE.MRD consortium is a group of experts, including scientists, technology, and pharmaceutical companies. The consortium is working on creating a reliable standard for the ctDNA tests, validating their clinical utility, and collecting data to help decide on the best treatment for each patient.

FRENCH.MRD.CRLM is the French study and part of the european GUIDE.MRD project.

DETAILED DESCRIPTION:
FRECNH.MRD.CRLM is a part of WP3 of the overarching GUIDE.MRD project. Each study chair has a local clinical trial protocol where patients are recruited. After the end of recruitment, samples will be analyzed under the GUIDE.MRD consortium.

The overall aim of GUIDE.MRD is to investigate the clinical utility of ctDNA analysis to predict and guide the choice of multi-modal therapies prospectively. The fundamental steps towards this aim are assessment and benchmarking of the many available ctDNA diagnostics to identify the best-suited tests for clinical application. Clinical samples will be used to benchmark ctDNA diagnostics and assess their true clinical performance. The samples should reflect clinical situations where the ctDNA diagnostics are particularly useful, such as post-operatively, post-adjuvant, during chemotherapy, and longitudinally during post-treatment surveillance. In these situations, ctDNA diagnostics could be used to either monitor treatment response (in case of MRD after surgery) or to identify relapse at an early time point. Based on ctDNA information, medical treatment could be changed, or radiology could be used to reveal the location of residual disease.

The rationale for the observational clinical study FRENCH.MRD.CRLM is to prospectively collect the clinical samples needed to enable assessment of the performance of ctDNA diagnostics in the setting of colorectal cancer (CRC). There are two main scenarios where ctDNA diagnostic is useful in CRC:

Metastatic CRC with isolated liver metastases. Metastatic CRC with liver metastases is a unique tumor type in that surgical resection or complete ablation of the metastases, is the standard of care. In virtually all other tumor types, resection of liver metastases is considered only within clinical trials or in exceptional clinical circumstances. In contrast, resection, or ablation of colorectal cancer liver metastases (CRLM) are routinely performed with curative intention, and the overall 5-year survival is around 50%. Most relapses present within three years after operative intervention. The clinical benefit of adjuvant chemotherapy is currently a matter of debate, due to limited data from randomized controlled trials and recent results that indicate inferior overall survival (OS) in patients who received adjuvant therapy (JCOG0603). Based on these and earlier data (EORTC Trial 40983) that failed to show an OS benefit of adjuvant therapy after CRLM resection, it can be assumed that most patients are treated unnecessarily with chemotherapy, and those patients that could receive targeted agents are missed. No histological or clinical markers are available to guide decisions on adjuvant treatment. In this setting, ctDNA could be valuable to guide decisions on adjuvant chemotherapy (yes/no), the addition of biologicals such as anti-VEGF and anti-EGFR agents, targeted therapies in the case of BRAF mutations, or the presence of microsatellite instability (MSI), for example.

PRIMARY OBJECTIVES Primary objective 1 (P1) To confirm that ctDNA analysis performed immediately after CRLM treatment can identify patients with a high risk of recurrence.

Specifically, the investigators want to determine the association between 3-year disease-free survival (DFS) and ctDNA detection status immediately after

1. Curative intended surgery and,
2. Postoperative chemotherapy.

SECONDARY OBJECTIVES Secondary objective 1 (S1) To technically assess, compare, and rank existing commercial ctDNA diagnostics after intended curative CRLM treatment (pre-operative chemotherapy, surgery or radiofrequency ablation +/- postoperative chemotherapy) to identify the best method at each time point, with no impact on diagnosis or treatment of patients enrolled in the study.

Secondary objective 2 (S2) To assess the effect of standard-of-care adjuvant chemotherapy on the level of ctDNA. Especially, for patients with ctDNA detected after surgery, the investigators will measure and compare the ctDNA levels in plasma samples drawn before and after adjuvant chemotherapy. Further, the change in ctDNA level will be correlated to the oncological outcomes (time to clinical recurrence, disease-free survival, and overall survival).

Secondary objective 3 (S3) To investigate if time to Molecular recurrence determined using serial ctDNA analyses in longitudinally collected plasma samples is shorter than time to Clinical recurrence using standard-of-care radiological imaging.

Secondary objective 4 (S4) To investigate the correlation between ctDNA analysis results and findings on CT scans. ctDNA analysis will be restricted to blood sampling times that are coinciding with standard-of-care CT scans during standard-ofcare surveillance. If ctDNA analysis can predict the outcome of the CT scan, the potential is that ctDNA analysis in the future can guide when to perform CT scans.

Secondary objective 5 (S5) To investigate the prognostic power of ctDNA at the time point of indeterminate CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older.
* Colorectal cancer liver metastasis or metastases, according to the assessment of the MDT.
* Metachronous and synchronous metastases will be included, as long as treatment intention of metastases resection is curative. In case of rare instances, where the liver metastases is removed before surgery of the primary tumor, postOP ctDNA is collected when the patient is considered completely tumor-free, i.e. after complete surgery of both the liver metastases and the primary tumor.
* Treatment is planned with curative intent (patients treated with RFA can be included, BUT in these cases a tissue sample from the primary CRC tumor is a requisite)

Exclusion Criteria:

* Hereditary colorectal cancer linked to familial colonic polyposis or Lynch syndrome.
* Extrahepatic metastases
* Malignant colorectal polyps diagnosed after polypectomy.
* Synchronous colorectal and non-colorectal cancer diagnosed per operative (except skin cancer other than melanoma)
* Other cancers (excluding colorectal cancer or skin cancer other than melanoma) within 3 years from eligibility screening
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude), inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study.
* Liver cirrhosis
* CRLM intervention/surgery cannot be/was not performed with curative intent
* No tumor tissue available (preferably CRLM lesion, or alternatively primary tumor)
* Pregnant or nursing woman, or in childbearing age and not willing to use contraception
* Protected and vulnerable adult
* Not covered by Health insurance
* Patient unable to understand and sign written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resectable colorectal liver metastasis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 3-year after the end of inclusion
  Disease-free survival was defined as the time between the date of the baseline blood sampling/inclusion and the date of the first event among or recurrence or death from any cause.

SECONDARY OUTCOMES:
Sensitivity (Se) of the ctDNA diagnostics | 3 years after the end of inclusion
  Sensitivity (Se) of the ctDNA diagnostics is calculated in subjects with a 3-year recurrence: Se = TP/(TP+FN) (a positive reference test)
Specificity (Sp) of the ctDNA diagnostics | 3 years after the end of inclusion
  Specificity (Sp) of the ctDNA diagnostics is calculated in subjects without a 3-year recurrence: Sp = TN/(TN+FP) (a negative reference test)
Positive predictive value of the ctDNA diagnostics | 3 years after the end of inclusion
  The predictive value of a positive test or positive predictive value (PPV): PPV = TP/(TP+FP).
Negative predictive value of the ctDNA diagnostics | 3 years after the end of inclusion
  The predictive value of a negative test or negative predictive value (NPV): NPV =TN/(TN+FN).
Area under the curve of the ctDNA diagnostics | 3 years after the end of inclusion
  Area Under the Curve of the of the ctDNA:
  * AUC ≤0.75 = low classification accuracy,
  * 0.75 < AUC < 0.85 = moderate accuracy,
  * and AUC ≥0.85 = high accuracy
Time to clinical recurrence | 3 years after the end of inclusion
  Time to clinical recurrence was defined as the time between the date of the baseline blood sampling/inclusion [debut] and the date of the recurrence.
Overall survival | 3 years after the end of inclusion
  Overall survival was defined as the time between the date of the baseline blood sampling/inclusion [debut] and the date of death from any cause.
Time to molecular recurrence | 3 years after the end of inclusion
  Time to molecular recurrence was defined as the time between the date of the baseline blood sampling/inclusion [debut] and the date of the molecular recurrence (positive ctDNA test).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BARDOL, M.D., Principal Investigator — University Hospital, Montpellier; Catherine ALIX-PANABIERES, Ph.D., Study Director — University Hospital, Montpellier